CLINICAL TRIAL: NCT02686164
Title: An Open-Label Phase 1 Study to Determine the Effect of Lenvatinib (E7080) on the Pharmacokinetics of Midazolam, a CYP3A4 Substrate, in Subjects With Advanced Solid Tumors
Brief Title: Phase 1 Study to Determine the Effect of Lenvatinib (E7080) on the Pharmacokinetics of Midazolam in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-A001-109
Record Dates: First submitted 2016-02-12; First posted 2016-02-19 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2018-01

CONDITIONS: Tumors
Keywords: Lenvatinib; Lenvima; E7080; Phase 1; Solid tumors; Midazolam; CYP3A4
MeSH Terms: conditions — Neoplasms | interventions — lenvatinib; Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- Lenvatinib + midazolam (Experimental): Participants with histologically confirmed unresectable or refractory solid tumors.
  Interventions: Drug: Lenvatinib; Drug: Midazolam

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib 24 mg (as one 4 mg and two 10 mg capsules) will be administered orally once daily with 240 mL (8 fluid oz) of water each morning, starting on Cycle 1 Day 1, in 28-day cycles.
  Other Names: Lenvima, E7080
Drug: Midazolam — Midazolam syrup 4 mg will be administered orally after an overnight fast on Cycle 1 Day -3 and concurrently with lenvatinib on Day 1 and Day 14 of Cycle 1. Participants will have to remain fasting for 2 hours after each dose of midazolam.

SUMMARY:
This is a multicenter, open-label, non-randomized Phase 1 study in participants with advanced solid tumors, excluding hepatocellular carcinoma (HCC), that have progressed after treatment with approved therapies, or for which there are no standard therapies available. The study will also include participants with radioiodine-refractory differentiated thyroid cancer (RR-DTC). Its primary intent is to determine the effect of lenvatinib on CYP3A4 activity as well as to assess the safety and activity of lenvatinib in these participants. The study will be conducted in the following 3 phases: Pretreatment Phase, Treatment Phase, and Extension Phase.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years at the time of informed consent.
2. Histologically or cytologically confirmed advanced solid tumors (excluding HCC) that have progressed following standard therapy, or for which no standard therapy exists (including surgery or radiation therapy) or participants with RR-DTC.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
4. Life expectancy greater than or equal to 3 months.
5. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP less than or equal to 150/90 mmHg at screening and no change in antihypertensive medications within 1 week prior to the Cycle 1 Day 1.
6. Adequate renal function defined as calculated creatinine clearance greater than or equal to 30 mL/min per the Cockcroft and Gault formula.
7. Adequate bone marrow function:

   1. Absolute neutrophil count (ANC) greater than or equal to 750/mm3 (greater than or equal to 0.75 X 10^9/L)
   2. Platelets greater than or equal to 75,000/mm3 (greater than or equal to 75 X 10^9/L)
   3. Hemoglobin greater than or equal to 9.0 g/dL
8. Adequate blood coagulation function as evidenced by an International Normalized Ratio (INR) less than or equal to 1.5.
9. Adequate liver function:

   1. Total bilirubin less than or equal to 1.5 X the upper limit of normal (ULN) except for unconjugated hyperbilirubinemia of Gilbert's syndrome
   2. Alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 X ULN (less than or equal to 5 X ULN if participant has liver metastases). If ALP is greater than 3 X ULN (in the absence of liver metastases) or greater than 5 X ULN (in the presence of liver metastases) AND the participant also is known to have bone metastases, the liver-specific ALP must be separated from the total and used to assess the liver function instead of total ALP.
10. Participants with Hepatitis B or C are eligible on the condition that they have adequate liver function as defined by Inclusion Criterion 9.
11. All prior therapy related toxicities must have resolved to Grade less than 2 severity per Common Terminology Criteria for Adverse Events (CTCAE version 4.03), except alopecia and infertility.
12. Left ventricular ejection fraction (LVEF) greater than 50% on echocardiography or multiple gated acquisition (MUGA) scan.
13. Females must not be lactating or pregnant at screening or baseline (as documented by a negative beta-human chorionic gonadotropin [B-hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of B-hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
14. Participant must voluntarily agree to provide written informed consent.
15. Participant must be willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

1. Participants with diagnosis of HCC.
2. Participants with anaplastic thyroid carcinoma with major blood vessel invasion or infiltration.
3. Participants having greater than (>) 1 plus (+) proteinuria on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with urine protein greater than or equal to (>=1) gram per 24 hours will be ineligible.
4. Participants with known leptomeningeal metastases or untreated brain metastases. Participants with known brain metastases will be eligible if they have completed the primary brain therapy (such as whole brain radiotherapy, stereotactic radiosurgery, or complete surgical resection) and if they have remained clinically stable, asymptomatic, and off steroids for at least 28 days.
5. Participants taking medications that are known potent CYP3A4 inducers/inhibitors or substrates with narrow therapeutic indices or St. John's Wort.
6. Participants unwilling to exclude grapefruit juice and grapefruit from their diet.
7. Participants who have received any anticancer treatment within 3 weeks or any investigational agent within 30 days before the first dose of study drug or who have not recovered from any acute toxicity greater than Grade 0 or 1 related to previous anticancer treatment.
8. Major surgery within 4 weeks before the first dose of study drug.
9. Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (eg, nausea, diarrhea, or vomiting) that might impair the bioavailability of lenvatinib or midazolam.
10. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of study drug; or cardiac arrhythmia requiring medical treatment (including oral anticoagulation).
11. A clinically significant electrocardiogram (ECG) abnormality (ie, corrected QT interval [QTc] interval greater than 480 msec when electrolyte balance is normal), or a history of risk factors for torsade de pointes, hypokalemia, long QT syndrome, or the use of concomitant medications resulting in a prolongation of QTc interval.
12. Active hemoptysis (bright red blood of at least 2.5 mL ie, half teaspoon) within 3 weeks prior to the first dose of study drug.
13. Active infection (any infection requiring treatment).
14. Known hypersensitivity to any component of lenvatinib or midazolam.
15. Prior treatment with lenvatinib.
16. Achlorhydria or use of antacids, proton-pump inhibitors, or other drugs known to raise gastric pH within 2 weeks before study drug administration.
17. Immunocompromised participants, including participants known to be infected with human immunodeficiency virus (HIV).
18. Any other major illness that, in the investigator's judgment, will substantially increase the risk associated with the participant's participation in this study.
19. Participants who meet any of the following criteria will be excluded from this study:

Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 international units per liter (IU/L) or equivalent units of ß-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.

OR Females of childbearing potential who do not agree to use a highly effective method of contraception for the entire study period and for 28 days after study drug discontinuation i.e. i) total abstinence (if it is their preferred and usual lifestyle) ii) an intrauterine device (IUD) or hormone releasing system (IUS) iii) a contraceptive implant iv. an oral contraceptive (with additional barrier method) OR who do not have a vasectomized partner with confirmed azoospermia. For sites outside of the European Union (EU), it is permissible that if a highly effective method of contraception is not appropriate or acceptable to the participant, then the participant must agree to use a medically acceptable method of contraception, i.e. double barrier methods of contraception such as condom plus diaphragm or cervical/vault cap with spermicide. All females will be considered to be of childbearing potential unless they are postmenopausal [amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause] or have been sterilized surgically [i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2018-08-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Facility # 1, Detroit, Michigan
  - Facility # 1, The Bronx, New York
  - Facility # 1, Philadelphia, Pennsylvania
  - Facility # 1, San Antonio, Texas

REFERENCES:
- [Derived] Shumaker R, Ren M, Aluri J, Dutcus CE, Rance C, He C. An Open-Label Phase 1 Study to Determine the Effect of Lenvatinib on the Pharmacokinetics of Midazolam, a CYP3A4 Substrate, in Patients with Advanced Solid Tumors. Eur J Drug Metab Pharmacokinet. 2020 Jun;45(3):373-383. doi: 10.1007/s13318-020-00607-7. PMID 32067158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in the United States from 18 Apr 2016 to 16 Aug 2018.
Pre-assignment Details: A total of 51 participants were screened and enrolled, of which 21 were screen failures and 30 participants received the study treatment.
Groups:
- Midazolam + Lenvatinib: Participants received midazolam 4 milligram (mg) (2 milliliter [mL]) syrup, orally, once daily (QD), after an overnight fast on Day -3, Day 1 and Day 14 of Cycle 1 and lenvatinib 24 mg capsules, orally, QD, on each morning, continuously for 28 days of Cycle 1, starting on Day 1 of Cycle 1. Participants continued to fast for 2 hours postdose of midazolam. Duration of each cycle equal to (=) 28 days.
Period: Overall Study
Arm/Group | Midazolam + Lenvatinib
Started | 30
Completed | 27
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal of consent | 1
Not completed — Clinical progression | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included participants who received at least 1 dose of midazolam or lenvatinib and had at least 1 postdose safety assessment.
Groups:
- Midazolam + Lenvatinib: Participants received midazolam 4 mg (2 mL) syrup, orally, QD, after an overnight fast on Day -3, Day 1 and Day 14 of Cycle 1 and lenvatinib 24 mg capsules, orally, QD, on each morning, continuously for 28 days of Cycle 1, starting on Day 1 of Cycle 1. Participants continued to fast for 2 hours postdose of midazolam. Duration of each cycle = 28 days.
Arm/Group | Midazolam + Lenvatinib
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (12.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 19
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-24): Area Under the Concentration-time Curve From Time Zero to 24 Hours Postdose for Midazolam and 1'-Hydroxymidazolam
Time Frame: Cycle 1 Day-3: 0-24 hours; Cycle 1 Day 1: 0-24 hours; Cycle 1 Day 14: 0-24 hours (Duration of each cycle=28 days)
Population: Pharmacokinetic (PK) analysis set included participants who had sufficient PK data to derive at least 1 PK parameter. Here number analyzed "n" are the participants who were evaluable for this outcome measure for given categories.
Measure: Mean (Standard Deviation); unit: hour*nanograms per milliliter (h*ng/mL)
Groups:
- Cycle 1 Day -3: Midazolam: Participants received midazolam 4 mg (2 mL) syrup, orally, QD, after an overnight fast on Day-3 of Cycle 1. Participants continued to fast for 2 hours post dose of midazolam.
- Cycle 1 Day 1: Lenvatinib + Midazolam: Participants received lenvatinib 24 mg capsules, orally, QD, in the morning and midazolam 4 mg (2 mL) syrup, orally, QD, after an overnight fast on Day 1 of Cycle 1. Participants continued to fast for 2 hours post dose of midazolam.
- Cycle 1 Day 14: Lenvatinib + Midazolam: Participants received lenvatinib 24 mg capsules, orally, QD, in the morning and midazolam 4 mg (2 mL) syrup, orally, QD, after an overnight fast on Day 14 of Cycle 1. Participants continued to fast for 2 hours post dose of midazolam.
Arm/Group | Cycle 1 Day -3: Midazolam | Cycle 1 Day 1: Lenvatinib + Midazolam | Cycle 1 Day 14: Lenvatinib + Midazolam
Number analyzed (Participants) | 29 | 29 | 29
hour*nanograms per milliliter (h*ng/mL)
  Midazolam: number analyzed (Participants) | 29 | 27 | 19
  Midazolam | 92.5 (34.5) | 89.7 (42.0) | 117 (61.1)
  1'-hydroxymidazolam: number analyzed (Participants) | 23 | 22 | 29
  1'-hydroxymidazolam | 38.5 (26.5) | 48.6 (47.8) | 41.3 (34.3)
Statistical Analysis 1: Comparison: Cycle 1 Day -3: Midazolam vs Cycle 1 Day 1: Lenvatinib + Midazolam; AUC(0-24) of Midazolam: Cycle 1 Day 1, Lenvatinib (single-dose) + Midazolam Versus (vs.) Cycle 1 Day -3, Midazolam; Test type: Other; Geometric Mean Ratio = 0.914, 90% CI 2-sided [0.850 to 0.983]
Statistical Analysis 2: Comparison: Cycle 1 Day -3: Midazolam vs Cycle 1 Day 14: Lenvatinib + Midazolam; AUC(0-24) of Midazolam: Cycle 1 Day 14, Lenvatinib (steady state) + Midazolam vs. Cycle 1 Day -3, Midazolam; Test type: Other; Geometric Mean Ratio = 1.148, 90% CI 2-sided [0.938 to 1.404]
Statistical Analysis 3: Comparison: Cycle 1 Day -3: Midazolam vs Cycle 1 Day 1: Lenvatinib + Midazolam; AUC(0-24) of 1'-hydroxy midazolam: Cycle 1 Day 1, Lenvatinib (single-dose) + Midazolam vs. Cycle 1 Day -3, Midazolam; Test type: Other; Geometric Mean Ratio = 1.120, 90% CI 2-sided [0.940 to 1.335]
Statistical Analysis 4: Comparison: Cycle 1 Day -3: Midazolam vs Cycle 1 Day 14: Lenvatinib + Midazolam; AUC(0-24) of 1'-hydroxy midazolam: Cycle 1 Day 14, Lenvatinib (steady-state) + Midazolam vs.Cycle 1 Day -3, Midazolam; Test type: Other; Geometric Mean Ratio = 1.199, 90% CI 2-sided [1.057 to 1.360]

2. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Midazolam and 1'-Hydroxymidazolam
Time Frame: Cycle 1 Day-3: 0-24 hours; Cycle 1 Day 1: 0-24 hours; Cycle 1 Day 14: 0-24 hours (Duration of each cycle=28 days)
Population: PK analysis set included participants who had sufficient PK data to derive at least 1 PK parameter. Here number analyzed "n" are the participants who were evaluable for this outcome measure for given categories.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cycle 1 Day -3: Midazolam | Cycle 1 Day 1: Lenvatinib + Midazolam | Cycle 1 Day 14: Lenvatinib + Midazolam
Number analyzed (Participants) | 29 | 29 | 29
nanogram per milliliter (ng/mL)
  Midazolam: number analyzed (Participants) | 29 | 28 | 19
  Midazolam | 26.5 (10.7) | 24.8 (17.4) | 28.3 (13.9)
  1'-hydroxy midazolam: number analyzed (Participants) | 29 | 28 | 19
  1'-hydroxy midazolam | 11.0 (8.64) | 12.7 (11.6) | 10.7 (11.6)
Statistical Analysis 1: Comparison: Cycle 1 Day -3: Midazolam vs Cycle 1 Day 1: Lenvatinib + Midazolam; Cmax of Midazolam: Cycle 1 Day 1, Lenvatinib (single-dose) + Midazolam vs. Cycle 1 Day -3, Midazolam; Test type: Other; Geometric Mean Ratio = 0.862, 90% CI 2-sided [0.753 to 0.988]
Statistical Analysis 2: Comparison: Cycle 1 Day -3: Midazolam vs Cycle 1 Day 14: Lenvatinib + Midazolam; Cmax of Midazolam: Cycle 1 Day 14, Lenvatinib (steady state) + Midazolam vs. Cycle 1 Day -3, Midazolam; Test type: Other; Geometric Mean Ratio = 1.027, 90% CI 2-sided [0.852 to 1.238]
Statistical Analysis 3: Comparison: Cycle 1 Day -3: Midazolam vs Cycle 1 Day 1: Lenvatinib + Midazolam; Cmax of 1'-hydroxy midazolam: Cycle 1 Day 1, Lenvatinib (single-dose) + Midazolam vs. Cycle 1 Day -3, Midazolam; Test type: Other; Geometric Mean Ratio = 1.055, 90% CI 2-sided [0.879 to 1.268]
Statistical Analysis 4: Comparison: Cycle 1 Day -3: Midazolam vs Cycle 1 Day 14: Lenvatinib + Midazolam; Cmax of 1'-hydroxy midazolam: Cycle 1 Day 14, Lenvatinib (steady state) + Midazolam vs. Cycle 1 Day -3, Midazolam; Test type: Other; Geometric Mean Ratio = 0.940, 90% CI 2-sided [0.845 to 1.046]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: First dose of study drug (Baseline) up to 28 days after last dose of study drug or until resolution, whichever came first (up to approximately 2.5 years)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Midazolam + Lenvatinib
Number analyzed (Participants) | 30
participants
  TEAEs | 30
  SAEs | 10

ADVERSE EVENTS:
Time Frame: First dose of study drug (Baseline) up to 28 days after last dose of study drug or until resolution, whichever came first (up to approximately 2.5 years)
Arm/Group | Midazolam + Lenvatinib
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 10/30
Other Adverse Events (participants affected / at risk) | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Midazolam + Lenvatinib (N=30)
Bradycardia (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Pyrexia (General disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Breast discharge (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Midazolam + Lenvatinib (N=30)
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Hypothyroidism (Endocrine disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 10
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 5
Chills (General disorders) | 3
Fatigue (General disorders) | 13
Oedema peripheral (General disorders) | 4
Urinary tract infection (Infections and infestations) | 2
Blood creatinine increased (Investigations) | 3
Weight decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No